CLINICAL TRIAL: NCT01592266
Title: F18-FLT PET/CT as a Tool for Assessment of Myeloablative Treatment in Patients With AML
Brief Title: F18-FLT PET/CT as a Tool for Assessment of Myeloablative Treatment in Patients With Acute Myeloid Leucemia(AML)
Acronym: AML F18-FLT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0112-12-HMO
Record Dates: First submitted 2012-04-16; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myeloid Leucemia
Keywords: FLT; PET; bone marrow; AML

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AML: patients with AML prior and after treatment

SUMMARY:
PET/CT is reliable tool in evaluation of treatment response in number cancers. F18-FLT is a precursor of DNA with high uptake in the bone marrow as a part of normal biodistribution. Highly increased uptake of this radiopharmaceutical was shown in a number of hematologic disease either in bone marrow or extramedullary.

F18-FLT PET/CT can provide a tool for whole body assessment of activity in bone marrow as well as early estimation of treatment efficacy or lack of it. In addition, this noninvasive study can replace bone marrow biopsy and predict response vs. non response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of AML

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with new diagnosis of AML
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Measure of extent and intensity ( by standardized uptake value - SUV) of disease in bone marrow demonstrated on PET/CT images before and after treatment.

SECONDARY OUTCOMES:
prediction of treatment response by dynamics of FLT uptake(by SUV)in comparison to bone marrow biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel